CLINICAL TRIAL: NCT01267331
Title: A Prospective,Randomized, Placebo-Controlled Study of Intramyocardial Injection of Autologous Bone-Marrow Mononuclear Cells in Patients With Severe, Chronic Ischemic Heart Disease Undergoing Coronary Bypass Surgery
Brief Title: Cell Therapy in Patients With Chronic Ischemic Heart Disease Undergoing Cardiac Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Gao Changqing, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006AA02A104
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2010-12

CONDITIONS: Old Myocardial Infarction; Chronic Myocardial Ischemia; Left Ventricular Dysfunction
Keywords: Old Myocardial Infarction; Stem Cell Therapy; Coronary Artery Bypass Grafting; Coronary Artery Disease
MeSH Terms: conditions — Ventricular Dysfunction, Left; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- stem cells injection (Experimental): Direct intramyocardial injection of autologous bone marrow mononuclear cells during CABG
  Interventions: Procedure: bone marrow mononuclear cells injection
- palcebo intramyocardial injection (Placebo Comparator): Direct intramyocardial injection of placebo containing saline and 5% human serum albumin during CABG.
  Interventions: Procedure: placebo intramyocardial injection

INTERVENTIONS:
Procedure: bone marrow mononuclear cells injection — Participants will receive direct intramyocardial injection of autologous bone marrow mononuclear cells during CABG.
  Other Names: autologous bone marrow mononuclear cells
  Arms: stem cells injection
Procedure: placebo intramyocardial injection — Participants will receive between 10 and 15 placebo injections that consist of saline and 5% human serum albumin during CABG.
  Other Names: palcebo
  Arms: palcebo intramyocardial injection

SUMMARY:
This prospective, randomized, placebo-controlled study was designed to assess the safety, feasibility and efficacy of intramyocardial injection of autologous bone marrow mononuclear cells in patients with severe, chronic ischemic disease scheduled to coronary artery bypass surgery.

DETAILED DESCRIPTION:
Severe ischemic heart disease remains a clinical challenge; many patients have undergone surgical myocardial revascularization procedures, but still remain symptomatic despite optimal medical therapy. Cell therapy with autologous bone marrow-derived cells (BMC) is a novel therapeutic strategy being tested for surgical treatment in patients with severe, chronic ischemic heart disease.

This research study is being performed to find out more information about the safety, feasibility, and efficacy of direct intramyocardial injection of autologous BMC on the myocardial perfusion and left ventricular function as an adjunctive therapy (compared to placebo) in patients undergoing coronary artery bypass surgery (CABG). The heart function evaluations will be performed by electrocardiogram, echocardiogram, and cMRI at baseline and during 6 months follow-up.

The secondary objective of this study is to assess the effect of intramyocardial injection of autologous BMC on functional class (angina/heart failure), global and cardiovascular mortality, and major adverse cardiac events after undergoing coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years.
2. Scheduled to undergo CABG.
3. At least 3 months since last episode of myocardial infarction.
4. Echocardiogram-assessed LVEF between 15 and 40% (Simpson's rule).
5. Abnormal wall motion of at least one segment due to prior myocardial infarction shown by echocardiography or left ventriculography.
6. Abnormal myocardial perfusion in infarcted area by SPECT.
7. Willingness to participate and ability to provide written informed consent.

Exclusion Criteria:

1. Contraindications to magnetic resonance imaging.
2. Need for urgent or emergent revascularization.
3. Severe valvular heart disease.
4. Confirmed myocardial infarction within 14 days, and/or rising cardiac biomarker proteins (i.e. troponin), and/or worsening ECG changes.
5. Prior cardiac surgery.
6. Stroke within 3 months prior to CABG.
7. Immunosuppressive medication (e.g. prednisone, cyclophosphamide, etanercept, etc.)
8. Severe chronic renal insufficiency (serum creatinine ≥ 200 mmol/dl or need for dialysis), liver disease, (diagnosis of cirrhosis, chronic hepatitis, or elevation of serum transaminases ≥3 times the upper limit of normal), cerebrovascular disease requiring concomitant carotid endarterectomy, peripheral arterial disease (claudication as the primary factor limiting activity), active non-dermatological malignancy requiring on-going treatment, or any other condition that would place the patient at increased risk for complications in the judgment of the attending cardiologist or cardiac surgeon
9. Hemoglobin less than 10g/dL, white blood cell count less than 4,000/mm3, absolute neutrophil count less than 1500/mm3
10. Active infection, with a temperature greater than 37.5°C within 48 hrs prior to surgery and an unexplained white blood cell count in excess of 10,000/mm3
11. Significant cognitive impairment.
12. Any condition associated with a life expectancy of less than 6 months.
13. Participation in other studies.
14. Positive laboratory test results for HIV, HBC, and HCV.
15. Pregnant woman.
16. Inability or unwillingness to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiac events | 6 months
  Freedom from Major Adverse Cardiac Event: cardiac death, myocardial infarction, repeat coronary bypass grafting or percutaneous intervention of bypassed artery

SECONDARY OUTCOMES:
left ventricular function | 6 months
  Globlal function,regional myocardial perfusion and function assessed by magnetic resonance iamge and echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Gao Changqing, MD, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China